CLINICAL TRIAL: NCT00995982
Title: VRC 309: A Multi-Center, Open-Label, Randomized Phase I Study of an Investigational Influenza DNA Vaccine Followed by 2009/2010 Seasonal Influenza Trivalent Inactivated Vaccine (TIV) Compared to Two Injections of TIV in Adults 45-70 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: RCHSPB
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100004; 10-I-0004
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-03

CONDITIONS: Influenza, Human
Keywords: Influenza; Healthy; Immunity; Preventive; Flu; HV; Healthy Volunteer
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: VRC-FLUDNA056-00VP

SUMMARY:
Background:

* Vaccines are substances used to try to create resistance or immunity to a disease and to prevent an infection. Investigators are looking into improved ways to give and test the results of different kinds of vaccines.
* Researchers are interested in comparing the results of an experimental DNA vaccine for the prevention of seasonal influenza against a standard FDA-approved vaccine for the prevention of seasonal influenza. The experimental DNA vaccine is not yet approved by the FDA for preventing the flu.

Objectives:

- To test the safety and immune response of an experimental DNA vaccine for seasonal influenza, compared to the standard vaccine for seasonal influenza.

Eligibility:

- Healthy individuals between ages 45 and 70 who have not yet received the seasonal influenza vaccine.

Design:

* Participants will have six planned clinic visits (Weeks 0, 1, 3, 4, 6, and 27) and two telephone follow-up contacts (within 2 days after each injection) during this study.
* Participants will be divided into two groups: one group will receive two standard (TIV) flu vaccine injections given using a needle and syringe, while the other will receive the DNA flu vaccine using a needleless injection system followed by the TIV vaccine.
* The vaccine injections for both groups will be given approximately 3 weeks apart,
* Clinic staff will observe participants for at least 30 minutes after each vaccination. One to two days after each injection, participants must telephone the clinic staff, and for 7 days after the vaccination participants will keep a diary card to report on possible side effects.
* During study visits, blood samples will be collected for research purposes to test for responses to vaccine.

DETAILED DESCRIPTION:
Study Design:

This is a Phase I, open-label study in healthy adults. The study will evaluate the safety, tolerability, and immunogenicity of a prime-boost vaccination regimen against the seasonal influenza virus with one dose of an investigational plasmid DNA vaccine as a prime followed 3 weeks later by the seasonal influenza trivalent inactivated vaccine (TIV) boost as compared to two injections with seasonal TIV. The hypothesis is that the DNA vaccine will be safe for administration and that the DNA vaccine prime - TIV boost schedule will elicit a greater frequency and/or magnitude of the antibody response than two injections with the seasonal TIV. The primary objective is to evaluate the safety and tolerability of the prime boost vaccine regimens. Secondary and exploratory objectives are related to evaluation of the major differences in quantity, quality and durability of humoral and cellular immune responses.

Product Description:

The VRC-FLUDNA056-00-VP vaccine was developed and manufactured by VRC, NIAID. It is composed of 3 closed-circular DNA plasmids, each with a CMV/R promoter, that encode for H1, H3, and influenza B hemagglutinin (HA) proteins from the same 2009-2010 influenza vaccine strains. DNA vaccine vials will be supplied at 4 mg/mL with each dose administered in a 1 mL volume. The TIV is the subunit inactivated vaccine for the 2009-2010 season. Each dose is composed of 45 microg hemagglutinin (HA) in 0.5 mL; with the recommended ratio of 15 microg HA of each of the following 3 strains: A/Brisbane/59/2007-like (H1N1); A/Brisbane/10/2007-like (H3N2); and B/Brisbane/60/2008-like. All injections will be administered intramuscularly (IM) in the deltoid muscle. The DNA injections will be administered by Biojector[Registered Trademark] 2000 Needle-Free Injection Management System and the TIV by needle and syringe.

Subjects:

60 healthy adults, 45-70 years old will be enrolled.

Study Plan:

There are two groups in the study randomized simultaneously at a ratio of 2:1 to the schedules shown in the schema. All subjects will receive the seasonal influenza TIV vaccine as the second injection.

The protocol requires 6 clinic visits (Weeks 0, 1, 3, 4, 6, 27) and 2 telephone follow-up contacts (within 2 days after each injection) for all groups.

ELIGIBILITY:
* INCLUSION CRITERIA:

A SUBJECT MUST MEET ALL OF THE FOLLOWING CRITERIA:

1. 45 to 70 years old.
2. Available for clinical follow-up through Week 27.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to donate blood for sample storage to be used for future research.
7. No evidence of previously undiagnosed clinically significant chronic diseases.
8. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) < 42 within the 56 days prior to enrollment.

   LABORATORY CRITERIA WITHIN 56 DAYS PRIOR TO ENROLLMENT:
9. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men
10. White blood cells (WBC) equal to 3,300-12,000 cells/mm(3)
11. Differential either within institutional normal range or accompanied by site physician approval as a differential that is consistent with healthy volunteer status
12. Total lymphocyte count greater than or equal to 800 cells/mm(3)
13. Platelets equal to 125,000 - 500,000/mm(3)
14. Alanine aminotransferase (ALT) less than or equal to 2.5 times upper limit of normal (ULN)
15. Serum creatinine less than or equal to 1 times ULN (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males).
16. Negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study].

    FEMALE-SPECIFIC CRITERIA:
17. Negative human chorionic gonadotropin (Beta-HCG) pregnancy test (urine or serum) for women presumed to be of reproductive potential on the day of enrollment.
18. A female subject must meet one of the following criteria:

    * No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

-Agrees to be heterosexually inactive at least 21 days prior to enrollment and through the last study visit,

OR

* Agrees to consistently practice contraception at least 21 days prior to enrollment and through the last study visit by one of the following methods:
* condoms, male or female, with or without a spermicide;
* diaphragm or cervical cap with spermicide;
* intrauterine device;
* contraceptive pills, patch, implant or any other FDA-approved contraceptive method;
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply:

Women Specific:

1. Breast-feeding or planning to become pregnant during the 27 weeks after enrollment in the study.

   Subject has received any of the following substances:
2. Seasonal influenza TIV within the 12 weeks prior to enrollment.
3. Systemic immunosuppressive medications or cytotoxic medications within the 12 weeks prior to enrollment. [With the exceptions that a short course (duration of 10 days or less or a single injection) of corticosteroids for a self-limited condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]
4. Blood products within 112 days (16 weeks) prior to HIV screening
5. Immunoglobulin within 56 days (8 weeks) prior to HIV screening
6. Live attenuated vaccines within 28 days (4 weeks) prior to initial study vaccine administration
7. Investigational research agents within 28 days (4 weeks) prior to initial study vaccine administration
8. Medically indicated subunit or killed vaccines (e.g., pneumococcal, or allergy treatment with antigen injections) within 14 days (2 weeks) of initial study vaccine administration
9. Current anti-TB prophylaxis or therapy

   Subject has a history of any of the following clinically significant conditions:
10. Contraindication to receiving an FDA approved current seasonal influenza vaccination (e.g., egg allergy).
11. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by investigator.
12. Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
13. Asthma that is severe, unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral, intravenous or high dose inhaled corticosteroids.
14. Diabetes mellitus type I.
15. Thyroid disease that is not well-controlled.
16. Generalized idiopathic urticaria within the last 1 year.
17. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
18. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
20. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Guillain-Barre Syndrome.
23. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt.
24. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10-08; Primary Completion 2010-09-03 (Actual); Study Completion 2010-09-03 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Clinical Alliance for Research and Education, Annandale, Virginia

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Luke CJ, Subbarao K. Vaccines for pandemic influenza. Emerg Infect Dis. 2006 Jan;12(1):66-72. doi: 10.3201/eid1201.051147. PMID 16494720
- [Background] Fiore AE, Shay DK, Broder K, Iskander JK, Uyeki TM, Mootrey G, Bresee JS, Cox NJ; Centers for Disease Control and Prevention. Prevention and control of seasonal influenza with vaccines: recommendations of the Advisory Committee on Immunization Practices (ACIP), 2009. MMWR Recomm Rep. 2009 Jul 31;58(RR-8):1-52. PMID 19644442
- [Derived] Ledgerwood JE, Hu Z, Costner P, Yamshchikov G, Enama ME, Plummer S, Hendel CS, Holman L, Larkin B, Gordon I, Bailer RT, Poretz DM, Sarwar U, Kabadi A, Koup R, Mascola JR, Graham BS; VRC 307 and VRC 309 Study Teams. Phase I clinical evaluation of seasonal influenza hemagglutinin (HA) DNA vaccine prime followed by trivalent influenza inactivated vaccine (IIV3) boost. Contemp Clin Trials. 2015 Sep;44:112-118. doi: 10.1016/j.cct.2015.08.006. Epub 2015 Aug 12. PMID 26275339